CLINICAL TRIAL: NCT03610308
Title: European Society for Trauma and Emergency Surgery (ESTES) Cohort Study Snapshot Audit 2018 - Acute Complicated Biliary Disease
Brief Title: ESTES Snapshot Audit 2018
Status: Completed | Type: Observational
Sponsor: European Society for Trauma and Emergency Surgery (Other)
Responsible Party: Principal Investigator, Gary Alan Bass, Chair, Emergency Surgery Cohort Studies Steering Group, European Society for Trauma and Emergency Surgery
Other Study IDs: ESTESSnapshotAudit2018
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Cholangitis; Gallstone; Pancreatitis Gallstone; Cholecystitis; Gangrenous
MeSH Terms: conditions — Cholangitis; Gallstones; Cholecystitis; Gangrene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore differences in patients, techniques and outcomes across the international cohort to identify areas of practice variability in the presentation and management of acute complicated calculous biliary disease.

DETAILED DESCRIPTION:
Background: Acute complications of biliary calculi are common, morbid and complex to manage. Variability exists in the techniques utilised to treat these conditions at a surgeon and unit level. This high-quality pan-European prospective audit will establish current practices and correlate them against outcomes.

Aim: To explore differences in patients, techniques and outcomes across the international cohort to identify areas of practice variability in the presentation and management of acute complicated calculous biliary disease.

Endpoints: A two-stage data collection strategy collecting patient demographics, details of operative, endocopic and radiologic intervention and outcome metrics. Several outcomes measures will be used including mortality, surgical morbidity (including Clavien-Dindo Grade 3a and above), ICU stay and length of hospital stay.

Methods: This 30 day prospective audit will be performed across Europe in late autumn 2018, and will be co-ordinated by the Emergency Surgery Cohort Study committee of European Society of Trauma and Emergency Surgery. This will be preceded by a one-week, three-centre pilot. Sites will be asked to pre-register for the audit and will be required to obtain appropriate regional or national approvals in advance of the enrolment date. The ESTES cohort studies committee will assist sites to register where possible.

During the study period, all eligible patients with acute complicated biliary calculous disease will be recorded contemporaneously and followed-up through to 60 days from their admission. The audit will be performed using a standardised pre-determined protocol and a secure online database. The report of this audit will be prepared in accordance with guidelines set by the STROBE (strengthening the reporting of observational studies in epidemiology) statement for observational studies.

Discussion: This multicentre, pan-European audit of acute complicated biliary calculous disease will be delivered by emergency surgeons and trainees in an organised and homogenous manner. The data obtained about areas of variability in provision or practice, and how this may impact upon outcomes, will serve to improve overall patient care as well as being hypothesis generating and inform areas needing future prospective study.

ELIGIBILITY:
* Inclusion Criteria:

  * Adult patients (over 18 years of age) admitted for:

    * Acute gangrenous or perforated calculous cholecystitis (AAST Severity Grade II or above)
    * Choledocholithiasis or complications of cholelithiasis and/or choledocholithiasis
    * Biliary Pancreatitis
* Procedures which should be included:

  1. Cholecystectomy (open, laparoscopic or robotic)
  2. Choledochotomy/common bile duct exploration (open, laparoscopic or robotic)
  3. Pancreatic necrosectomy
  4. Gastrojejunostomy
  5. Cyst gastrostomy
  6. Endoscopic retrograde choledochopancreatography (ERCP) or Endoscopic ultrasound (EUS)
  7. Percutaneous cholecystostomy (transhepatic or transperitoneal)
  8. Percutaneous transhepatic drainage, stone removal or stent placement
* Exclusion Criteria:

  * Uncomplicated biliary colic
  * Biliary dyskinesia
  * Acute calculous cholecystitis (AAST Grade I)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Pan-European, prospective audit of consecutive patients admitted for the treatment of complicated calculous biliary disease over a 30-day study period. The audit shall include unscheduled admissions from 1 October 2018 to 31 October 2018.
  * Commencement timeframe: The sites will start within a time window from 1 October to 31 October 2018. Following commencement, the sites will be required to include all eligible consecutive patients for 30 consecutive days.
  * Final date for operation inclusion: The sites can include admissions that occur up to 31 October 2018.
  * All patients will be followed for 60 days post-admission. Data collection should therefore be completed by 31 December 2018.
  * As this is an observational cohort audit, no change to normal patient management is required.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 60 days
  Overall and disease-related mortality

SECONDARY OUTCOMES:
ICU Admission | 60 days
  Intensive Care Unit admission for organ-supportive therapy
Length of hospital stay | 60 days
  Length of hospital stay
Complications | 60 days
  Complication related to surgical, endoscopic or radiologic intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gary A Bass, MD, MSc, MBA, Study Chair — Tallaght University Hospital, Dublin, Ireland; Shahin Mohseni, MD, PhD, Principal Investigator — Örebro University Hospital, Sweden; Jorge Pereira, MD, FACS, Principal Investigator — Hospital de São Teotónio, Viseu, Portugal; Amy Gillis, MD, MCh, FRCSC, Principal Investigator — Tallaght University Hospital, Dublin, Ireland
Locations (1):
- Tallaght University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bass GA, Gillis AE, Cao Y, Mohseni S; European Society for Trauma and Emergency Surgery (ESTES) Cohort Studies Group. Patients over 65 years with Acute Complicated Calculous Biliary Disease are Treated Differently-Results and Insights from the ESTES Snapshot Audit. World J Surg. 2021 Jul;45(7):2046-2055. doi: 10.1007/s00268-021-06052-0. Epub 2021 Apr 3. PMID 33813631